CLINICAL TRIAL: NCT00703430
Title: The Effect of Memantine on Aggression and Agitation and Its Impact on Caregiver Burden of Patients With Alzheimer's Disease: A 12-week Open-label Study
Brief Title: Memantine on Aggression and Agitation of Alzheimer's Disease (AD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Principal Investigator, Xin Yu, Institute Director, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CN-IIT-12292
Record Dates: First submitted 2008-06-20; First posted 2008-06-23 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease, agitation, aggression, dementia
MeSH Terms: conditions — Alzheimer Disease; Psychomotor Agitation; Aggression; Dementia | interventions — Memantine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Memantine
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Memantine — Initially Memantine 5mg/day, titrated within the first month to a maintenance dose of 20mg/day, which is maintained for the following 2 months.
  Other Names: Ebixa®

SUMMARY:
Alzheimer's disease (AD), is associated with behavioral disturbances in approximately 50% of AD patients in Beijing. Agitation, and aggression specifically, is considered the most serious noncognitive symptom experienced in patients with dementia. Memantine is a recognized treatment for Alzheimer's disease either alone or in combination with cholinesterase inhibitors. Its efficacy in vascular dementia is also established. Family members continue to play a central role in home care for the demented elderly in China. This proposal is to conduct a study in Beijing, China to investigate the efficacy and safety of Memantine in the treatment of agitation and aggression in AD patients. In addition, this proposal aims to explore the impact of memantine on caregiver burden of AD patients in Chinese culture.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Clinical diagnosis of Alzheimer's disease.
3. Having at least a minimum aggression score on the Cohen-Mansfield Agitation Inventory (CMAI): a score of ≥ 4 on at least 1 aggressive item, or a score of 3 on at least 2 aggressive items, or a score of 2 on at least 3 aggressive items, or 2 aggressive items occurring at a frequency of 2 and 1 at a frequency of 3.
4. Availability of a responsible family member or carer to ensure treatment compliance and provide information for informant assessments.

Exclusion Criteria:

1. Unavailability of a responsible family member or carer
2. Severe renal impairment.
3. History of seizures
4. Diagnosis of any concomitant life threatening illness.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-03; Primary Completion 2013-12 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
CMAI score | 12 weeks

SECONDARY OUTCOMES:
CBI score | 12 weeks
RUD | 12 weeks
NPI score | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xin Yu, MD, Principal Investigator — Peking University Institute of Mental Health
Locations (1):
- Peking University Institute of Mental Health, Beijing, China